CLINICAL TRIAL: NCT04139967
Title: Prospective Study of Short Course Radiation Therapy for Elderly Patients With Rectal Cancer
Brief Title: Study of Short Course Radiation Therapy for Elderly Patients With Rectal Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: recruitment rates were too low
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Haoming (Carl) Qiu, Associate Professor, University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4297
Record Dates: First submitted 2019-10-23; First posted 2019-10-25 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Cancer, Rectal
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Elderly rectal cancer patients (Experimental)
  Interventions: Radiation: Short course radiation therapy

INTERVENTIONS:
Radiation: Short course radiation therapy — 25 Gray in 5 fractions over 5-7 days

SUMMARY:
This study will help determine if a short course of radiation therapy is effective to treat rectal cancer in older patients. A shorter course of radiation treatment may be better tolerated than a longer course or surgery for the treatment of rectal cancer in the elderly.

ELIGIBILITY:
Inclusion Criteria:

* 70 years or older at time of diagnosis
* No restrictions on gender or ethnicity
* Ability and willingness to make follow up appointments
* Pathologic diagnosis of rectal cancer
* Presentation could be symptomatic or asymptomatic
* T1-T3 primary rectal adenocarcinoma as determined on TRUS, CT, or MRI pelvis
* Peri-rectal node positive allowed
* Inability to tolerate radical surgery, as judged by geriatric oncology or surgeon and tumor board OR patient refusal of surgery
* Inability to receive chemoradiation therapy, defined as concurrent chemotherapy and radiation doses of 45-50.4 Gy, as judged by radiation, medical, or geriatric oncology
* Patients with dementia eligible if Health Care Proxy (HCP) is available and supportive of follow up schedule

Exclusion Criteria:

* Age under 70 years of age
* Ability and desire to receive definitive surgical intervention
* Ability and desire to receive concurrent chemoradiation therapy

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 2 (Actual)
Dates: Start 2020-01-20 (Actual); Primary Completion 2022-08-03 (Actual); Study Completion 2022-08-03 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | 5 years
  Progression will be defined as Radiologic response from MRI or CT scans using RECIST v1.1 criteria.
Number of participants who experience a grade 2 adverse event | week 5
  CTCAE V4.0 will be used to determine the grade 2 AE.

SECONDARY OUTCOMES:
Number of participants who received surgery for their cancer | 5 years
Number of participant who experience metastatic disease | 5 years
  MRI or endoscopy will be used to track metastasis to other parts of the body
Change in Mean quality of life | baseline to 24 months
  Quality of life will be assessed using the Low Anterior Resection Syndrome Score Questionnaire. Scores range from 0-42 points with higher scores indicating worse outcome.
Change in Mean functional status | baseline to 24 months
  Quality of life will be assessed using the Low Anterior Resection Syndrome Score Questionnaire. Scores range from 0-42 points with higher scores indicating worse outcome.
Number of participants with improved symptoms | 5 years
  Symptoms will be documented by the treating physician at each clinical visit for 5 years.

CONTACTS AND LOCATIONS:
Locations (1):
- James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No